CLINICAL TRIAL: NCT01565291
Title: A Preliminary Evaluation of the Amyloid Binding Properties, Pharmacokinetics and Safety of 18F-AV-45 in Healthy Elderly Volunteers and Patients With Alzheimer's Disease
Brief Title: A Preliminary Study of 18F-AV-45 in Alzheimer's Disease and Healthy Elderly Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A01
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects With AD (Experimental): Probable AD, National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, with mild/moderate dementia (Mini-Mental State Examination (MMSE) from 10 to 24)
  Interventions: Drug: florbetapir F 18
- Healthy Elderly Subjects (Experimental): Cognitively normal with MMSE of 29 or higher; age 50 years or older
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
A preliminary study to test how florbetapir F 18 (18F-AV-45) acts in the brains and bodies of healthy elderly people and patients with Alzheimer's Disease (AD) by using a positron emission tomography (PET) scanner.

ELIGIBILITY:
Inclusion Criteria (AD group):

* Probable AD according to the National Institute of Neurological and Communication Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Mild/moderate dementia as evidenced by a mini mental state exam (MMSE) score ranging from 10 to 24, boundaries included, at screening
* History of cognitive decline had been gradual in onset and progressive over a period of at least 6 months

Inclusion Criteria (healthy volunteer group):

* No evidence of significant cognitive impairment by history and psychometric testing
* MMSE of 29 or higher

Exclusion Criteria (both groups):

* Neurodegenerative disorders other than AD
* Cognitive impairment resulting from trauma, hypoxic damage, vitamin deficiency, brain infection, brain cancer, endocrine disease, or mental retardation
* Clinically significant infarct or possible multi-infarct dementia as defined by the NINCDS criteria
* Evidence on screening MRI or other biomarker that suggests alternate etiology for cognitive deficit (for healthy controls, evidence suggesting the presence of AD pathology)
* Clinically significant psychiatric disease
* History of epilepsy or convulsions
* Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Current clinically significant cardiovascular disease
* Received investigational medication within the last 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (3):
- United States (3):
  - Research Site, Baltimore, Maryland
  - Research Site, North East, Maryland
  - Research Site, Long Branch, New Jersey

REFERENCES:
- [Result] Wong DF, Rosenberg PB, Zhou Y, Kumar A, Raymont V, Ravert HT, Dannals RF, Nandi A, Brasic JR, Ye W, Hilton J, Lyketsos C, Kung HF, Joshi AD, Skovronsky DM, Pontecorvo MJ. In vivo imaging of amyloid deposition in Alzheimer disease using the radioligand 18F-AV-45 (florbetapir [corrected] F 18). J Nucl Med. 2010 Jun;51(6):913-20. doi: 10.2967/jnumed.109.069088. PMID 20501908

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With AD: Probable AD, National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, with mild/moderate dementia (Mini-Mental State Examination [MMSE] from 10 to 24)
Period: Overall Study
Arm/Group | Subjects With AD | Healthy Elderly Subjects
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With AD | Healthy Elderly Subjects | Total
Number analyzed (Participants) | 16 | 16 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 75.8 (9.2) | 72.5 (11.56) | 74.3 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Cortical to Cerebellum SUVR
Description: Standardized Uptake Value ratio (SUVR) is the ratio of tracer uptake in predefined cortical regions, relative to uptake in the cerebellum gray matter. Total scan length was 200 min.
Time Frame: 50-60 min after injection
Population: 4 subjects in AD group and 1 subject in the healthy elderly group were excluded due to poor placement and/or excessive movement in the scanner during the 200-minute procedure.
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Subjects With AD | Healthy Elderly Subjects
Number analyzed (Participants) | 11 | 15
SUVR | 1.665 (0.175) | 1.246 (0.177)

2. Secondary Outcome: Precuneus to Cerebellum SUVR
Description: Ratio of uptake in the precuneus to uptake in the cerebellum.
Time Frame: 50-60 min after injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Subjects With AD | Healthy Elderly Subjects
Number analyzed (Participants) | 11 | 15
SUVR | 1.847 (0.237) | 1.300 (0.271)

ADVERSE EVENTS:
Time Frame: AEs occuring within 3 days of injection. SAEs occuring within 30 days of injection
Arm/Group | Subjects With AD | Healthy Elderly Subjects
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With AD (N=16) | Healthy Elderly Subjects (N=16)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
CLAUSTROPHOBIA (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days